CLINICAL TRIAL: NCT07305311
Title: Characterising the Network-Specific Effects of Piriform Cortex Stimulation Via SEEG With Multimodal Data Integration
Brief Title: Characterising the Network-Specific Effects of Piriform Cortex Stimulation Via SEEG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-292-202
Record Dates: First submitted 2025-12-02; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Refractory Epilepsy; Neuromodulation
Keywords: SEEG; Piriform cortex; Electrical stimulation; Electrophysiology
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SEEG recordings and SPES effects (Experimental): This arm encompasses patients with drug-resistant focal epilepsy who underwent intracranial monitoring via stereotactically implanted depth electrodes (SEEG) as part of their standard presurgical evaluation. During the monitoring period, these patients additionally underwent systematic Single-Pulse Electrical Stimulation (SPES) mapping. SPES was administered according to a standardized clinical protocol, involving the delivery of single, low-intensity electrical pulses to selected electrode contacts-including those located within or adjacent to the piriform cortex-while recording the evoked electrophysiological responses across the implanted SEEG network. The data collected in this arm include continuous intracranial EEG recordings, precise stimulation parameters (location, intensity), and the corresponding electrophysiological responses used to characterize cortico-cortical evoked potentials and network connectivity.
  Interventions: Device: SEEG recordings and SPES

INTERVENTIONS:
Device: SEEG recordings and SPES — The intervention involves single-pulse electrical stimulation (SPES) applied during stereotactic electroencephalography (SEEG) monitoring. Low-intensity, standardized electrical pulses are delivered to targeted contacts within or near the piriform cortex via implanted depth electrodes, while simultaneous full-bandwidth SEEG recordings capture network-wide electrophysiological responses, allowing characterization of stimulation-evoked brain network activation and modulation patterns.

SUMMARY:
The prospective study aims to characterize the network-specific modulatory effects of piriform cortex stimulation in patients undergoing stereotactic EEG for drug-resistant epilepsy. Using multimodal data, it seeks to link stimulation-evoked electrophysiological responses across brain networks with clinical outcomes, to inform targeted neuromodulation therapies.

DETAILED DESCRIPTION:
This study employs stereotactic electroencephalography (SEEG) to investigate the network-specific mechanisms of brain modulation induced by electrical stimulation of the piriform cortex. By analyzing high-density intracranial recordings, combined with structural and functional neuroimaging, the research systematically characterizes how focal stimulation differentially engages and reorganizes activity across large-scale neural circuits. The primary focus is to decode the electrophysiological signatures of network engagement-including changes in spectral power, phase synchronization, and information flow-to reveal fundamental principles of targeted neuromodulation in the human brain.

ELIGIBILITY:
Inclusion Criteria:

* The patients were diagnosed with drug-resistant epilepsy.
* The patients underwent stereoelectroencephalography (SEEG) implantation for pre-surgical evaluation of epilepsy, with at least one electrode target reaching the piriform cortex
* Participants/parents/legal guardian provide informed consent for inclusion

Exclusion Criteria:

* Subjects that experience surgical complications during the implant procedure will be excluded from the study

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2027-01-08 (Estimated); Study Completion 2027-11-08 (Estimated)

PRIMARY OUTCOMES:
Seizure Discharge Suppression Rate | 72 hours
  Quantified as the percentage reduction in the frequency of spikes and interictal epileptiform discharges (IEDs) during active stimulation compared to the baseline period.

SECONDARY OUTCOMES:
Single-Pulse Stimulation Amplitude: | 72 hours
  The minimum current intensity (mA) required to elicit a reproducible response.
N1 Component Amplitude and Latency: | 72 hours
  Amplitude (μV) and latency (ms) of the primary cortical evoked response (N1 wave).
Spatial Distribution of Activation | 72 hours
  The extent of cortical activation, assessed by the number of electrode contacts showing significant evoked responses.
Effective Connectivity Change： | 72 hours
  Alterations in effective connectivity strength (e.g., measured by Granger causality within a 500 ms time window).
Phase-Amplitude Coupling Index | 72 hours
  Changes in coupling between the phase of low-frequency oscillations and the amplitude of the gamma band (30-80 Hz).
Functional Network Reconfiguration | 72 hours
  Changes in node centrality metrics (e.g., betweenness centrality, degree centrality) based on graph-theoretical analysis of functional networks.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 72 hours
  Adverse Events: Incidence and severity of adverse events specifically associated with piriform cortex stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No